CLINICAL TRIAL: NCT05015738
Title: Digital Tools for Learning Diabetes: Combination of Animation and Gamification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Ayse Kabuk, RN, PhD, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: University of Health Sciences
Record Dates: First submitted 2021-08-06; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Diabetes; Educational Problems
Keywords: diabetes; distance learning; digital tools; gamification; animation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study was conducted between Octorber and November 2020 on 70 volunteer students studying in the Department of Nursing at the Faculty of Health Sciences in Turkey. The inclusion criteria were as follows: (a) being 18 years old or over, (b) studying in the second year, (c) volunteering to take a diabetes course (d) not attending any course for diabetes before e) have a smart phone f) no internet connection problem g) not to be absent on the date when the data of the research will be collected. The second-year nursing students were selected for the study since they have not taken diabetes courses before. The students included in the study were randomly divided into two groups.The control group was taught with the traditional method and the experimental group was taught with learning activities based on animation and gamification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional diabetes education (Other): The subjects and activities were applied to the control group, who received traditional diabetes education, between 8:00 and 10:00 with the classical method, which lasted 2 hours, for 10 weeks. The training was completed by the researcher with the verbal narration method. "Diabetes Achievement Assessment Test" with question and answer method was administered to the students at the beginning and end of the application. These questions were the same questions asked to the experimental group. Interaction of groups with each other was limited. Students were informed about this and their consent was taken.At the end of the course, students' opinions were taken through the form developed by the researchers. Instructional Materials Motivation Survey (IMMS) was used to measure to student' motivation levels.
  Interventions: Other: Traditional education
- Diabetes Education supported by digital tools (Experimental): The subjects included in the course content were given between 10:00-12:00 with the animation supported method, which lasted for 2 hours. The animations were created by the researchers to reflect all guidelines for diabetes. The scenario of the animation video was prepared in line with the training content. Storyboards in videos and animations were created with the collaboration of researchers and experts in their fields (software specialists, computer programmers). The animation video was voiced in Turkish by a professional actor. Animations are 2 minutes each and a total of 18 minutes long. The 'Kahoot' application, a Web 2.0 tool, was used to apply Diabetes Achievement Evaluation Test. At the end of the course, students' opinions were taken through the form developed by the researchers. Instructional Materials Motivation Survey (IMMS) was used to measure to student' motivation levels.
  Interventions: Device: Diabetes Education supported by digital tools

INTERVENTIONS:
Other: Traditional education — Diabetes education will be given by the trainer for 10 weeks, 2 hours of presentation.
  Arms: Traditional diabetes education
Device: Diabetes Education supported by digital tools — Diabetes education will be given for 10 weeks with 2-minute animations. At the end of the course, learners' knowledge was measured with a knowledge test using the Kahoot app.
  Arms: Diabetes Education supported by digital tools

SUMMARY:
COVID-19, a global epidemic that affects the world, has created significant changes in many areas, especially in the health system. One of the most affected areas is nursing education. The content of nursing education focuses on cognitive, psychomotor and affective areas. In order for nursing education to be successful, important initiatives should be provided in the education of these areas. However, difficulties were encountered in the distance education process.

This study was conducted to evaluate the delivery of diabetes education in nursing with animation and gamification.

DETAILED DESCRIPTION:
This study was conducted with a randomized-controlled experimental design. This study was conducted between October and November 2020 in the Department of Nursing at the Faculty of Health Sciences in Turkey. The inclusion criteria were as follows: being 18 years old or over, studying in the second year, volunteering to take a diabetes course, not attending any course for diabetes before, have a remote access tool (internet connection, personel comuter eg.), not to be absent on the date when the data of the research will be collected. The second-year nursing students were selected for the study since participants have not taken diabetes nursing courses before.

In the randomization part of the study, the students were assigned to the experiment (n=35) and control (n=35) groups according to their number in the class list using the random numbers table.

Data were callacted with "Structured Student Identification Form", "Diabete Nursing Knowledge Test", "Instructional Materials Motivation Survey" and " Opinion Form on Diabetes Education Program supported by digital tools".

The Diabetes Nursing course is 2 hours per week fow 10 week. After students were assigned to groups with randomization, the application process of the research was explained to the students. The control group was taught with the traditional method and the experimental group was taught with learning activities based on animation and gamification.

Direct lecture, question-answer teaching methods were used through Microsoft Power Point presentation to the control group of Diabetes Nursing course. At the end of the lesson, "Diabete Nursing Knowledge Test" and "Instructional Materials Motivation Survey" were used in control group.

An animated video was watched at the beginning of each lesson in the experimental group. Later, lecture and question-answer teaching methods were used through Microsoft Power Point presentation. At the end of each lesson, Web 2.0 (Kahoot) application was used to reinforce students' knowledge.At the end of the lesson, "Diabete Nursing Knowledge Test", "Instructional Materials Motivation Survey" and " Opinion Form on Diabetes Education Program supported by digital tools"were used in intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Over18 years old
* Being 2nd year student
* Volunteering to take a diabetes course
* Not attending any course for diabetes before
* Have a remote access tool (internet connection, personel comuter eg.)
* Not to be absent on the date when the data of the research will be collected.

Exclusion Criteria:

* Not being volunteer to participate in the study
* who have taken the course in previous years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Diabetes Nursing Course Knowledge Test, 10. week (after the course finished) | Through study completion, an average of 3 mounth
  This knowledge test, which is prepared by submitting to expert opinion, consists of 40 multiple-choice questions. Each question is worth 2,5 points. The higher the test score, the higher the level of knowledge.
Instructional Materials Motivation Survey (IMMS), 10. week (after the course finished) | Through study completion, an average of 3 mounth
  The scale was prepared in a 5-point Likert type, 36 items. The highest score that can be obtained from the entire scale is 165, and the lowest score is 33. The increase in the score obtained from the scale is interpreted as an increase in the motivation towards the teaching material.

SECONDARY OUTCOMES:
Opinion Form on Diabetes Education Program supported by digital tools, for only experimental group, 10. week (at the end of the course) | Through study completion, an average of 3 mounth
  The form was prepared for the students in the experimental group to determine their views on education supported by animation and gamification. IThe form consisted of 4 open-ended questions containing opinions and suggestions about teaching method and digital education materials.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Kabuk, Dr, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If it is necessary for the ethical issue, we can share.

REFERENCES:
- [Background] Liaw SY, Wong LF, Chan SW, Ho JT, Mordiffi SZ, Ang SB, Goh PS, Ang EN. Designing and evaluating an interactive multimedia Web-based simulation for developing nurses' competencies in acute nursing care: randomized controlled trial. J Med Internet Res. 2015 Jan 12;17(1):e5. doi: 10.2196/jmir.3853. PMID 25583029
- [Background] Du S, Liu Z, Liu S, Yin H, Xu G, Zhang H, Wang A. Web-based distance learning for nurse education: a systematic review. Int Nurs Rev. 2013 Jun;60(2):167-77. doi: 10.1111/inr.12015. Epub 2013 Mar 25. PMID 23691999
- [Background] Fayaz A, Mazahery A, Hosseinzadeh M, Yazdanpanah S. Video-based Learning Versus Traditional Method for Preclinical Course of Complete Denture Fabrication. J Dent (Shiraz). 2015 Mar;16(1 Suppl):21-8. PMID 26106631
- [Background] Koch J, Andrew S, Salamonson Y, Everett B, Davidson PM. Nursing students' perception of a Web-based intervention to support learning. Nurse Educ Today. 2010 Aug;30(6):584-90. doi: 10.1016/j.nedt.2009.12.005. Epub 2010 Jan 4. PMID 20045583
- See also: Federation of European Nurses in Diabetes — https://www.fend.org/